CLINICAL TRIAL: NCT01370668
Title: Comparative Efficacy of Two Psychosocial Strategies of Intervention (Neurocognitive vs Psychoeducative) as add-on Therapy Versus Treatment as Usual in Bipolar Disorder
Brief Title: Functional Remediation for Bipolar Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centro de Investigación Biomédica en Red de Salud Mental (Network)
Collaborators: Hospital Clinic of Barcelona (Other); Benito Menni (Unknown); University of Valencia (Other); Hospital Universitari de Bellvitge (Other); Universidad de Oviedo (Other); Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other); Hospital General Universitario Gregorio Marañon (Other); Hospital Santiago Apóstol de Vitoria (Unknown); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Eduard Vieta, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI08/90094; PI080180 (Other Grant/Funding Number: Fondo Investigaciones Sanitarias)
Record Dates: First submitted 2011-03-10; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Bipolar Disorder
Keywords: functional remediation; psychoeducation; neurocognition
MeSH Terms: conditions — Bipolar Disorder | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Functional remediation (Experimental): Patients assigned to the experimental treatment will receive standard psychiatric care and will be enrolled in the neurocognitive intervention program composed of 21 sessions of 90 minutes, each aimed at improving the following cognitive domains: attention, memory and executive functions and psychosocial functioning.
  The program will be performed in an 8-to-10 patient group conducted by 2 experienced neuropsychologists. with previous experience with bipolar patients (at least 3 years) and specific training on patients' group management.
  Interventions: Behavioral: Functional remediation
- Psychoeducation (Active Comparator): The group psychoeducation is a tested (Colom et al, 2003) and manualized intervention (Vieta and Colom, 2006) consisting on 21 sessions of 90 minutes, aimed at improving 4 main issues: illness awareness, treatment adherence, early detection of prodromal symptoms and recurrences and lifestyle regularity. The program will be performed in an 8-10 patient group conducted by 2 experienced psychologists with previous experience with bipolar patients and specific training on patients' group management. The structure of each session consists of a 30 to 40 minute speech on the topic of the day, followed by an exercise related to the issue (eg. drawing a life chart, writing a list of potential triggering factors) and a discussion.
  Interventions: Behavioral: Psychoeducation
- Treatment as Usual (Active Comparator): This arm will not receive any sort of add-on psychosocial intervention. All patients will keep on receiving standard psychiatric treatment.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: Functional remediation — The functional remediation program is composed of 21 weekly sessions of 90 minutes, each aimed at improving the following cognitive domains: attention, memory and executive functions and psychosocial functioning.
  The program will be performed in an 12- to 15-patient group conducted by 2 experienced neuropsychologists with previous experience with bipolar patients and specific training on patients' group management.
  Arms: Functional remediation
Behavioral: Psychoeducation — Group psychoeducation is a tested and manualized intervention consisting of 21 weekly sessions of 90 minutes aimed at improving 4 main issues: illness awareness, treatment adherence, early detection of prodromal symptoms and recurrences, and lifestyle regularity.
  Arms: Psychoeducation
Behavioral: Treatment as usual — The patients will not receive any add-on psychosocial intervention. All patients will keep on receiving standard psychiatric treatment.
  Arms: Treatment as Usual

SUMMARY:
Bipolar disorder is a severe, chronic and recurrent illness, that affects nearly the 5% of the population. Recent research point at the relevance and persistence of cognitive dysfunctions in bipolar patients even beyond the acute phases, although cognitive impairment has been classically associated with schizophrenia and not bipolar disorder. Current findings suggest that some intervention is needed in order to improve not only affective symptoms but also cognitive dysfunctions, so that patients could benefit from cognitive remediation techniques to improve cognitive impairment and the functional outcome. There is no previous research on the efficacy of cognitive remediation programs on bipolar disorder.

DETAILED DESCRIPTION:
The method consists of a randomized clinical trial with 3 arms: 1) one group (n=66) will receive a cognitive rehabilitation program + pharmacological treatment, 2) another group (n=66) will receive a psychoeducation program + pharmacological treatment, and 3) a control group (n=66) will only receive pharmacological treatment. A psychopathological, neuropsychological and functional assessment will be administered pre and post-intervention and a 12-month follow-up to assess the long term effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Diagnosis of bipolar disorder type I or II, according to DSM-IV-TR 4ª Ed criteria
* Adult patients, aged between 18 and 55 years old
* Euthymic (YMRS < 6, HDRS < 8) for at least three months prior to study entry.
* Signed inform consent
* Severe or moderate functional impairment (FAST > 18)

Exclusion Criteria:

* IQ < 85
* Neurological illness
* Present diagnosis of substance abuse or dependence according to DSM-IV criteria the last three months
* Significant medical illness considered as severe by the study that may interfere with assessments
* having been enrolled in any kind of cognitive rehabilitation intervention the last two years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 198 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Functional Assessment Short Test (FAST) | Baseline
  The FAST is a valid and reliable instrument, easy to apply which requires a short period of time to administer. Evaluates functioning taking into account the last 15 days. It was developed for the clinical evaluation of the main difficulties presented by psychiatric patients, and has been validated in several languages for patients with bipolar disorder. The FAST scale consists of 24 items which allow the assessment of six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time.
Functional Assessment Short Test (FAST) | 6 months
  The FAST is a valid and reliable instrument, easy to apply which requires a short period of time to administer. Evaluates functioning taking into account the last 15 days. It was developed for the clinical evaluation of the main difficulties presented by psychiatric patients, and has been validated in several languages for patients with bipolar disorder. The FAST scale consists of 24 items which allow the assessment of six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time.
Functional Assessment Short Test (FAST) | 12 months
  The FAST is a valid and reliable instrument, easy to apply which requires a short period of time to administer. Evaluates functioning taking into account the last 15 days. It was developed for the clinical evaluation of the main difficulties presented by psychiatric patients, and has been validated in several languages for patients with bipolar disorder. The FAST scale consists of 24 items which allow the assessment of six specific areas of functioning: autonomy, occupational functioning, cognitive functioning, financial issues, interpersonal relationships and leisure time.

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vieta, MD, PhD, Principal Investigator — Centro de Investigación Biomédica en Red de Salud Mental

REFERENCES:
- [Derived] Bonnin CM, Torrent C, Arango C, Amann BL, Sole B, Gonzalez-Pinto A, Crespo JM, Tabares-Seisdedos R, Reinares M, Ayuso-Mateos JL, Garcia-Portilla MP, Ibanez A, Salamero M, Vieta E, Martinez-Aran A; CIBERSAM Functional Remediation Group. Functional remediation in bipolar disorder: 1-year follow-up of neurocognitive and functional outcome. Br J Psychiatry. 2016 Jan;208(1):87-93. doi: 10.1192/bjp.bp.114.162123. Epub 2015 Nov 5. PMID 26541692
- [Derived] Sole B, Bonnin CM, Mayoral M, Amann BL, Torres I, Gonzalez-Pinto A, Jimenez E, Crespo JM, Colom F, Tabares-Seisdedos R, Reinares M, Ayuso-Mateos JL, Soria S, Garcia-Portilla MP, Ibanez A, Vieta E, Martinez-Aran A, Torrent C; CIBERSAM Functional Remediation Group. Functional remediation for patients with bipolar II disorder: improvement of functioning and subsyndromal symptoms. Eur Neuropsychopharmacol. 2015 Feb;25(2):257-64. doi: 10.1016/j.euroneuro.2014.05.010. Epub 2014 May 20. PMID 24906790
- [Derived] Torrent C, Bonnin Cdel M, Martinez-Aran A, Valle J, Amann BL, Gonzalez-Pinto A, Crespo JM, Ibanez A, Garcia-Portilla MP, Tabares-Seisdedos R, Arango C, Colom F, Sole B, Pacchiarotti I, Rosa AR, Ayuso-Mateos JL, Anaya C, Fernandez P, Landin-Romero R, Alonso-Lana S, Ortiz-Gil J, Segura B, Barbeito S, Vega P, Fernandez M, Ugarte A, Subira M, Cerrillo E, Custal N, Menchon JM, Saiz-Ruiz J, Rodao JM, Isella S, Alegria A, Al-Halabi S, Bobes J, Galvan G, Saiz PA, Balanza-Martinez V, Selva G, Fuentes-Dura I, Correa P, Mayoral M, Chiclana G, Merchan-Naranjo J, Rapado-Castro M, Salamero M, Vieta E. Efficacy of functional remediation in bipolar disorder: a multicenter randomized controlled study. Am J Psychiatry. 2013 Aug;170(8):852-9. doi: 10.1176/appi.ajp.2012.12070971. PMID 23511717